CLINICAL TRIAL: NCT01542918
Title: Lenalidomide Plus Rituximab for Recurrent/Refractory CNS and Intraocular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Rubenstein (Other)
Collaborators: Celgene (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, James Rubenstein, Associate Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112530; NCI-2013-00056 (Registry Identifier: Cancer Trial Reporting Program)
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Recurrent/Refractory CNS; Intraocular Lymphoma
Keywords: Recurrent; Refractory; CNS; Intraocular; Lymphoma
MeSH Terms: conditions — Recurrence; Intraocular Lymphoma; Lymphoma | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study intervention (Experimental): Lenalidomide Plus Rituximab
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Formulation of Dosage forms: 5 mg, 10 mg, 15 mg and 25 mg capsules.
  Dosage: 10 mg - 30 mg (Treatment 1 and Treatment 2)
  Route of administration: Oral
  Other Names: Revlimid
Drug: Rituximab — Formulation of Dosage forms: 100 mg/IO mL and 500 mg/50 mL solution in a single-use vial
  Dosage: 375 mg/m2, intravenous (Treatment 2, Cycle 1 only); 25 mg intraventricular injection (Treatment 2, all cycles)
  Route of administration: Intravenous (Treatment 2, Cycle 1 only); Intraventricular injection (Treatment 2, all cycles)
  Other Names: Rituxan; MabThera

SUMMARY:
This is a Phase I study, which means that the goal is to see if the study treatment is safe. The purpose of this study is to test the safety of Lenalidomide at different dose levels, and to test the safety of Lenalidomide alone or in combination with Rituximab (also known as Rituxan®).

DETAILED DESCRIPTION:
Rationale for the Proposed Study

There is evidence that immunomodulatory drugs such as lenalidomide stimulate immune effectors such as natural killer (NK) cells, and thus promote rituximab efficacy via ADCC. Because of the evidence for synergy between rituximab and lenalidomide in NHL, patients who do not respond to lenalidomide monotherapy will receive combined intravenous plus intraventricular rituximab in addition to lenalidomide. To maximize delivery to the central nervous system (CNS), the investigators propose to administer rituximab via both intravenous and intraventricular routes. The rationale for intraventricular administration of rituximab is the demonstration that approximately 0.1% of systemically administered rituximab penetrates the cerebral spinal fluid (CSF) but that intraventricular administration of rituximab is both feasible and achieves high concentrations that are associated with anti-lymphoma activity. This study will thus build upon the two Phase 1 trials of intraventricular rituximab that have been conducted at University of California, San Francisco (UCSF) to define the safety of the intraventricular route of administration; this study will, however, be the first to evaluate the combination of intraventricular plus intravenous treatment.

The rationale for intravenous administration of rituximab in recurrent CNS lymphoma is that the blood-brain-barrier is likely partially disrupted, particularly when there is lymphoma-associated contrast enhancement detectable on the MRI, and the fact that there is evidence for activity when rituximab is administered intravenously, both as monotherapy (Batchelor et al., 2011) and potentially in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent and willingness to comply with the requirements of the protocol
* Age eighteen years or older
* Tumors must be CD20+ on prior pathologic analysis
* All prospective participants must have an Ommaya reservoir (or equivalent ventricular access device) inserted as part of their standard clinical care prior to initiation of study treatment.
* No concurrent methotrexate, thiotepa, cytarabine, or investigational agents
* Absolute neutrophil count (ANC) > 1,500 (growth factors permitted)
* Platelets >50,000 (platelet transfusion allowed)
* Total bilirubin </= 1.5 x upper limit of normal (ULN)
* aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) </= 3 x ULN.
* Stable dose of glucocorticoids pre-therapy. If patients are receiving dexamethasone, the dose of dexamethasone should not increase during the 96 hours prior to initiation of therapy.
* Renal function assessed by calculated creatinine clearance. Patients must have calculated creatinine clearance (CrCl) >/= 60ml/min by Cockcroft-Gault formula or 24 hour urine demonstrating CrCl >/= 60ml/min .
* Females of childbearing potential (FCBPs)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 Milli-International Units per millilitre (mIU/mL) within 10 - 14 days and again within 24 hours prior to receiving lenalidomide for Cycle 1 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBPs must also agree to ongoing pregnancy testing and for 28 days after receiving their last dose of lenalidomide.
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin).
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

* Intraventricular chemotherapy or radiation therapy within 4 days of starting treatment
* Intravenous rituximab within 30 days of starting treatment
* Persistent neurotoxicity from intraventricular methotrexate, cytarabine, thiotepa
* Anticipated survival of less than 1 month
* Pregnant women and women of child-bearing potential who are not using an effective method of birth control.
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Contraindication to aspirin. If unable to take aspirin, contraindication to warfarin or low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
To establish the maximal tolerated dose (MTD) of Lenalidomide in patients with recurrent CNS NHL and intraocular NHL | Participants will be followed for the duration of treatment, an expected average of 4 months.

SECONDARY OUTCOMES:
To define the extent of cerebrospinal fluid (CSF) penetration of lenalidomide. | Participants will have CSF withdrawn every 4 weeks while on treatment. Average study participation is approximately 4 months.
To assess the clinical efficacy Lenalidomide monotherapy as measured by cytologic, neurologic, radiographic, and ocular (for patients with intraocular lymphoma) response criteria. | Participants will have weekly evaluations at clinic visits for the duration of treatment. Average study participation is approximately 4 months.
To define the immunological effects of lenalidomide using flow-cytometry CSF as well as genomic markers of recurrent/refractory CNS lymphoma. | Participants will have CSF withdrawn every 4 weeks while on treatment. Average study participation is approximately 4 months.
To assess the clinical efficacy of combined intraventricular plus systemic rituximab administration in combination with lenalidomide as measured by cytologic, neurologic, and radiographic response criteria. | Participants will have weekly evaluations at clinic visits for the duration of treatment. Average study participation is approximately 4 months.
  Objective only applies to patients with recurrent CNS lymphoma not responding to lenalidomide as monotherapy
To determine a potential impact of intravenous rituximab administration on the rate of rituximab clearance from the CSF after intraventricular rituximab administration. | Participants will have CSF withdrawn every 4 weeks while on treatment. Average study participation is approximately 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: James Rubenstein, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rubenstein JL, Geng H, Fraser EJ, Formaker P, Chen L, Sharma J, Killea P, Choi K, Ventura J, Kurhanewicz J, Lowell C, Hwang J, Treseler P, Sneed PK, Li J, Wang X, Chen N, Gangoiti J, Munster PN, Damato B. Phase 1 investigation of lenalidomide/rituximab plus outcomes of lenalidomide maintenance in relapsed CNS lymphoma. Blood Adv. 2018 Jul 10;2(13):1595-1607. doi: 10.1182/bloodadvances.2017014845. PMID 29986852